CLINICAL TRIAL: NCT02881606
Title: Evaluation of the Clinical Effectiveness of Naso-alveolar Molding (NAM) Versus Computer Aided Design NAM (CAD/NAM) in Infants With Bilateral Cleft Lip and Palate: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Ali El Ashmawi, Assistant lecturer at orthodontic department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2016-08-184
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Cleft Lip and Palate
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Blinding was done for the plastic surgeon (care provider) during lip repair and for the outcome assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naso-alveolar molding (NAM) (Active Comparator): Active plates and nasal stents (Grayson method)
  Interventions: Device: Naso-alveolar molding (NAM)
- Computer aided design NAM (CAD/NAM) (Active Comparator): Computer aided design active plates and nasal stents
  Interventions: Device: Computer aided design NAM (CAD/NAM)

INTERVENTIONS:
Device: Naso-alveolar molding (NAM)
  Arms: Naso-alveolar molding (NAM)
Device: Computer aided design NAM (CAD/NAM)
  Arms: Computer aided design NAM (CAD/NAM)

SUMMARY:
Bilateral cleft lip and palate neonates will be randomly assigned to one of two groups: (gp1 presurgical Naso-alveolar molding (NAM) using Grayson method, gp 2 computer aided design NAM (CAD/NAM). The aim of the study is to compare between short term clinical effects of both interventions as regards alveolar alignment, nasal esthetics and interlabial gap.

ELIGIBILITY:
Inclusion Criteria:

• Bilateral cleft lip and palate

Exclusion Criteria:

Patients without cleft palate Unilateral cleft lip Patients having systemic medical problems that contraindicate NAM treatment Patients with history of previous presurgical infant orthopedics Patients with history of any surgical procedures (ex: lip adhesion)

Ages: 7 Days to 60 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2016-12; Primary Completion 2019-03 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Alveolar alignment | 5-6 months
  Reference points,lines and planes on digital models recording the symmetry and alignment of maxillary arch segments

SECONDARY OUTCOMES:
Nasal and labial esthetics | 5-6 months
  Reference points, lines and planes on standardized photos recording the collumellar length, symmetry of nostrils and interlabial gap

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medicine, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol